CLINICAL TRIAL: NCT00668057
Title: Randomized, Double-blind, Multi-centre, Parallel-goup Study to Investigate the Efficacy and Safety of Three Doses of BAY38-9456 (5 mg, 10 mg and 20 mg) Versus Placebo in the Treatment of Patients With Erectile Dysfunction
Brief Title: BAY38-9456 (Vardenafil HCL Tablet) in ED Treatment for China Registration.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10690
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Erectile Dysfunction
Keywords: Male Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 3 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 5 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 6 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 5 mg Vardenafil orally 1 hour prior to sexual intercourse
  Arms: Arm 1
Drug: Levitra (Vardenafil, BAY38-9456) — 10 mg Vardenafil orally 1 hour prior to sexual intercourse
  Arms: Arm 2
Drug: Levitra (Vardenafil, BAY38-9456) — 20 mg Vardenafil orally 1 hour prior to sexual intercourse
  Arms: Arm 3
Drug: Placebo — 5 mg matching placebo
  Arms: Arm 4
Drug: Placebo — 10 mg matching placebo
  Arms: Arm 5
Drug: Placebo — 20 mg matching placebo
  Arms: Arm 6

SUMMARY:
This study was to compare the efficacy of 3 doses of vardenafil, 5 mg, 10 mg and 20 mg, with matching placebo in Chinese male ED patients, treated for a maximum of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men with ED for more than 6 months. ED defined according to the National Institute of Health, USA Department of Health and Human Services, consensus statement, as the inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance.
* Stable heterosexual relationship

Exclusion Criteria:

* Primary hypoactive sexual desire- History of myocardial infarction, stroke or life-threatening arrhythmia within the 6-month period prior to Visit 1 (Week -4)
* Nitrate use
* Other exclusion criteria apply

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2002-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Erectile Function domain score of the International Index of Erectile Function, questions 1-5 and 15 | 12 weeks

SECONDARY OUTCOMES:
Global Assessment Questionnaire | 12 weeks
Erectile Function domain score of the International Index of Erectile Function | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- China (3):
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai